CLINICAL TRIAL: NCT02665819
Title: SALTO-BIO (Long Term Follow up in Oncology) - PanCareLIFE. Long Term Support for Pediatric Cancer Survivors in Rhône-Alpes. Evaluation of Women Fertility.
Brief Title: Long Term Support for Pediatric Cancer Adult Survivors in Rhône-Alpes : Evaluation of Women Fertility.
Acronym: SALTO-BIO
Status: Completed | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Saint Etienne (Other)
Responsible Party: Sponsor
Other Study IDs: 1508057; 2015-A00667-42 (Other: ANSM)
Record Dates: First submitted 2016-01-25; First posted 2016-01-28 (Estimated); Last update posted 2018-02-20 (Actual); Status verified 2018-02

CONDITIONS: Pediatric Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — 25 ml of blood for each patient will be necessary to measure the AMH and FSH hormones rates.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Pediatric cancer women survivors: Women diagnosed for a cancer between 01/01/87 and 31/12/99 before the age of 15 years old living in Rhône-Alpes, will incur a blood taking for DNA tests (hormone tests) to see their fertility capacity.
  Interventions: Other: Pediatric cancer women survivors

INTERVENTIONS:
Other: Pediatric cancer women survivors — Women will incur a blood taking to obtain fertility indication.

SUMMARY:
PanCareLIFE Study is a cohort study of patients treated for cancer in childhood, and biological case-control study nested in the cohort (WP4) is coordinated by Erasmus MC-Sophia Children's Hospital in Holland.

Ensure optimal patient quality of life throughout his life is a priority for the research teams. PanCareLIFE Study also aims to identify the factors that predispose to impaired quality of life. It is in this light that will be offered to patients a quality of life questionnaires during the period of treatment and then periodically during long-term follow-up.

DETAILED DESCRIPTION:
PanCareLIFE Study is a cohort study of patients treated for cancer in childhood, and biological case-control study nested in the cohort (WP4) is coordinated by Erasmus MC-Sophia Children's Hospital in Holland. At European level, approximately 1,200 women are expected in this latest study, the patients were already identified through certain regional or national registries in terms of cumulative doses of chemotherapy, surgery, radiation.

Ensure optimal patient quality of life throughout his life is a priority for the research teams. PanCareLIFE Study also aims to identify the factors that predispose to impaired quality of life. It is in this light that will be offered to former patients to complete quality of life questionnaires during the period of treatment and then periodically during long-term follow-up.

The SALTO-BIO study is the French part of the European study PanCareLIFE. CHU of Saint-Etienne as French promotor, will organize this study only on the Rhône-Alpes region (Lyon, Grenoble and Saint-Etienne centers) and will participate as co-investigator and "data provider "to WP2, WP3, WP4 and WP6. Indeed, ototoxicity is already studied by a French group.

ELIGIBILITY:
Inclusion Criteria:

* min 18 years old
* female
* diagnosed for a cancer between 01/01/87 and 31/12/99, before 15 years old, and living in Rhône-Alpes
* treated with chemotherapy +/- radiotherapy
* accepting a blood taking to perform DNA and hormonal tests
* affiliated to a security social scheme
* informed consent

Exclusion Criteria:

- severe mental disorder

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The population studied belongs to a cohort composed of women treated for a cancer in their childhood (diagnosed between 1987 and 1999 in Rhône-Alpes Region) before 15 years old.
Sampling Method: Probability Sample
Enrollment: 101 (Actual)
Dates: Start 2015-10-23 (Actual); Primary Completion 2016-11-29 (Actual); Study Completion 2016-11-29 (Actual)

PRIMARY OUTCOMES:
Measure the FSH hormone rate. | Day 1
  In this arm women will incur a blood taking to measure the FSH hormone rate.
Measure the AMH hormone rate. | Day 1
  In this arm women will incur a blood taking to measure the AMH hormone rate.
Detect the genetic polymorphism of the FSH and AMH hormones. | Day 1
  With the blood taking realized for each patient, genetic markers will be obtained to identify their fertility capacity.

SECONDARY OUTCOMES:
Quality of life | Day 1
  The quality of life for each patient will be measured with the SF-36 scale.
Identification of new loci associated to ovarian toxicity | Day 1
  With a pan-genomic method, new loci (associated to ovarian toxicity) will be identified.

CONTACTS AND LOCATIONS:
Overall Officials: BERGER Claire, MD, Principal Investigator — CHU SAINT-ETIENNE; Léonie CASAGRANDA, PhD, Study Chair — CHU SAINT-ETIENNE
Locations (4):
- France (4):
  - Chu Grenoble, Grenoble
  - IHOP 1 Lyon, Lyon
  - CH Lyon Sud, Pierre-Bénite
  - CHU Saint-Etienne, Saint-Etienne

IPD SHARING:
Plan to Share IPD: No